CLINICAL TRIAL: NCT04078893
Title: The Effect of Recruiting Inactive Blood Donors Using Different Means : on "Need" or Just Keeping Communication
Brief Title: The Effect of Recruiting Inactive Blood Donors Using Different Means
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guangzhou Blood Center (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: recruit inactive blood donors
Record Dates: First submitted 2019-08-27; First posted 2019-09-06 (Actual); Last update posted 2019-10-21 (Actual); Status verified 2019-10

CONDITIONS: Blood Donors
Keywords: inactivated donors recruitment, on need ,communication

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- control group (No Intervention)
- on need group (Experimental)
  Interventions: Other: telephone recruitment
- communication group (Experimental)
  Interventions: Other: telephone recruitment

INTERVENTIONS:
Other: telephone recruitment — using telephone to recruit inactive donors on two different methods
  Arms: communication group; on need group

SUMMARY:
14098 inactive donors were randomly divided into three groups according to age, sex, blood donation frequency,time of last donation and blood donation site, one group acted as the control group, one will be recruited by telephone recruitment on "need", and one will just be called for improvement suggestions of blood donor service.

ELIGIBILITY:
Inclusion Criteria:

* inactive donors during 2016-2018

Exclusion Criteria:

* inactive donors during 2016-2018 but not eligible to donate

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14098 (Estimated)
Dates: Start 2019-10-20 (Estimated); Primary Completion 2019-11-29 (Estimated); Study Completion 2020-01-29 (Estimated)

PRIMARY OUTCOMES:
donate blood or not | 12 months
  rate of donation after recruitment

CONTACTS AND LOCATIONS:
Locations (1):
- Guangzhou Blood Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Yes
To compare the effect of recruiting inactive blood donors between on "need" and just keeping communication
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code